CLINICAL TRIAL: NCT05215977
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study, Evaluating the Efficacy and Safety of Recombinant Fully Human Anti-RANKL Monoclonal Antibody in Postmenopausal Osteoporosis Subjects With Increased Bone Fracture Risk
Brief Title: Efficacy and Safety of MW031 in PMO Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW031-2019-CP301
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MW031 (Experimental): MW031 injection(60 mg) was administered subcutaneously once every 6 months for a maximum of 2 consecutive doses throughout the trial, according to the investigator's assessment.
  Interventions: Drug: MW031
- placebo (Placebo Comparator): Placebo was administered subcutaneously once every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MW031 — The active ingredient of MW031 is a recombinant human anti-RANKL monoclonal antibody ,subcutaneous injection of 60 mg (1.0 mL)every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Dietary Supplement: Elemental Calcium Oral, at least1000 mg Dietary Supplement: Vitamin D Oral, 400 IU
  Other Names: Recombinant anti-RANKL human monoclonal antibody injection
  Arms: MW031
Drug: Placebo — subcutaneous injection of 60 mg (1.0 mL)every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Dietary Supplement: Elemental Calcium Oral, at least1000 mg Dietary Supplement: Vitamin D Oral, 400 IU
  Arms: placebo

SUMMARY:
This study is a multicenter, randomized, double-blinded, placebo-controlled Phase III clinical study to evaluate the clinical efficacy and safety of MW031 in Chinese postmenopausal osteoporotic subjects with increased bone fracture risk .

ELIGIBILITY:
Inclusion Criteria:

* BMD -4.0<T-score ≤-2.5 at either the lumbar spine or total hip or femoral neck
* All subjects must have at least one of following additional the risk factors:history of fracture, parental history of hip fracture, increased bone turnover rate at screening, low body weight, elderly (age≥65year)，current smoker
* Postmenopausal is defined as >2 years postmenopausal, which can be >2 years of spontaneous amenorrhea, or bilateral oophorectomy >2 years after surgery. If bilateral oophorectomy status is unknown, use follicle-stimulating hormone (FSH) levels > 40 mIU/mL to confirm surgical postmenopausal status.

Exclusion Criteria:

* Bone/metabolic disease
* Hyperparathyroidism or hypoparathyroidism
* Thyroid condition: Hyperthyroidism or hypothyroidism
* Rheumatoid arthritis
* Malignant tumors
* Malabsorption syndrome
* Oral bisphosphonates

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) at the Lumbar Spine from Baseline up to 12 months | Baseline and Month 12
  Dual energy x-ray absorptiometry (DXA) is applied for Bone mineral density (BMD) assessment.

SECONDARY OUTCOMES:
Percent Change in BMD at the Lumbar Spine from Baseline up to 6 months | Baseline and Month 6
Percent change in BMD at the total hip, femoral neck from Baseline up to 6 months and 12 months | Baseline, Month 6 and Month 12
Percent Change in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) and Serum Procollagen Type I N Propeptideserum (s-PINP) from Baseline up to 12 months | Baseline, Month 1, Month 3, Month 6, Month 9 and Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Y, Huo Y, Li Y, Kong X, Wang B, Liu F, Zheng X, Li Y, Yang Y, Xu Y, Xue Q, Hu Z, Xiao Y, Ma W, Guo Y, Yu W, Xia W. Randomized, double-blind, placebo-controlled, multicenter study to evaluate efficacy and safety of the denosumab biosimilar MW031 in Chinese postmenopausal women with osteoporosis. Expert Opin Biol Ther. 2024 Jul;24(7):665-672. doi: 10.1080/14712598.2024.2352587. Epub 2024 May 16. PMID 38752402